CLINICAL TRIAL: NCT06878677
Title: Individualized Exercise Prescription With a Data-driven Approach in Individuals With Stroke - A Feasible Study
Brief Title: Individualized Exercise Prescription With a Data-driven Approach in Individuals With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Patrick Kwong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20240216001
Record Dates: First submitted 2025-03-03; First posted 2025-03-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke Gait Rehabilitation; Stroke Patients; Stroke
Keywords: stroke; lower extremities; gait; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two arm randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Data-driven exercise group (Experimental): Based on the results of the gait patterns, the PI will design appropriate exercises that target the specific gait impairment at a specific time period during the gait cycle. Exercises will utilize various modalities that are commonly used in clinical practice, including TheraBand, gym equipment, free weight. The training may target single-joint movement or targeting a movement pattern that involves multiple joint holistically. A body harness system will be used to protect the participant during the exercise training. The participant will be supervised by a research assistant who has rich experience in conducting exercise training on people with disability.
  Interventions: Other: Data-driven exercise
- Standarzied exercise group (Placebo Comparator): Participants in the standard exercise group will undergo a standardised exercise programme consisting of five lower-limb exercises commonly employed in clinical settings and prescribed to patients as home exercises. They include (1) stepping up and down to strengthen the muscles of both legs and to improve control in shifting the center of gravity; (2) heel-raising exercises on an inclined wedge to strengthen both ankle plantarflexors; (3) assuming a semi-squatting position to improve lower-limb muscle endurance and proprioception in the knees and ankles; (4) standing on a dura disk to improve dynamic standing balance; (5) walking across obstacles to enhance anticipatory postural control.
  Interventions: Behavioral: Standardized exercises

INTERVENTIONS:
Other: Data-driven exercise — The result from the Statistical Parametric Mapping 1D (SPM1D) analysis will be used to identify the magnitude of deviation from normal gait patterns in reference to healthy subjects for each lower limb joint. Thereby, the targeted action and joint position can be identified. Training will focus on the specific movement where the "steepest gradients" are observed.
  The targeted exercises will be selected based on the five largest deviations observed during the swing or stance phase. Open-chain exercises will be applied to address deviations in the swing phase, while closed-chain exercises will be applied to address deviation in the stance phase. Each exercise will be performed for approximately 80-100 repetitions, with a total duration of 10 minutes per exercise, including rest periods.
  Arms: Data-driven exercise group
Behavioral: Standardized exercises — The participants will perform dose match standardised exericse program.
  Arms: Standarzied exercise group

SUMMARY:
The goal of this clinical trial is to evaluate if the exercised via data-driven approach is effective in enhance the gait pattern in people with stroke. It will reduce burdun of patient consultations for clinicians in reality.The main questions it aims to answer are:

Does individualized exercise training programmes via data-driven approach could improve gait patterns in individuals with chronic stroke? Does individualized exercise training programmes via data-driven approach could improve improve motor recovery, motor functions (including gait speed and balance performance), and community integration in individuals with chronic stroke?

Participants will:

Undergo 12 supervised-exercise (training sessions (60 minutes, two times a week, for six weeks), Participants will receive a data-driven exercise prescription or conventional exercise prescription which consists of 5 different exercises.

They will be assessed on Baseline assessment before training (A0); after six sessions (A1); after 12 sessions (A2); and three months after training (A3).

DETAILED DESCRIPTION:
Based on the results of the gait patterns and Electromyography (EMG) analysis, the principal investigator (PI) will design appropriate exercises that target the specific gait impairment at a specific time period during the gait cycle. Exercises will utilize various modalities that are commonly used in clinical practice, including TheraBand, gym equipment, free weight. The training may target single-joint movement or targeting a movement pattern that involves multiple joint holistically. A body harness system will be used to protect the participant during the exercise training. The participant will be supervised by a research assistant who has rich experience in conducting exercise training on people with disability. Below are potential exercises that will be prescribed to the participant based on their impairment revealed by the analyses. eg. Lack of hip flexion during swing phase: Open kinetic chain strengthing exercise for hip flexor in a concentric manner...

ELIGIBILITY:
Inclusion Criteria:

* between 45 and 75 years old;
* have received a diagnosis of stroke more than six months earlier;
* able to walk 10 m independently;
* able to score at least 6 of 10 on the Abbreviated Mental Test;
* able to follow instructions and give informed consent.

Exclusion Criteria:

* any existing medical condition such as uncontrolled hypertension that hindered training or assessment;
* unable to offer consent due to impaired cognitive function.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Gait kinematics | At baseline and 6 weeks post-intervention
  Seventeen wearable sensors (Inertial Measurement Units, IMUs) were attached to the participants' bodies in accordance with the Xsens user manual to collect kinematic data. The extracted data included the pelvis tilt angle (°), oblique angle (°), and rotation angle (°); hip flexion angle (°) and abduction angle (°); knee bending angle (°); as well as ankle flexion angle (°) and abduction angle (°), which were used for further analysis. These data were converted into standardized gait cycles (101 time points) for statistical parametric mapping (SPM1D) analysis, and the deviation time from the normal reference was compared to determine whether there were changes in deviation timing before and after the treatment.

SECONDARY OUTCOMES:
Electromyography (EMG) signals in Maximum Voluntary Contraction (MVC) and muscle activation during gait | At baseline and 6 weeks post-intervention
  Twelve Electromyography (EMG) sensors were placed on the left and right sides of the gluteus maximus, gluteus medius, quadriceps, hamstrings, tibialis anterior, and gastrocnemius muscles to measure Maximum Voluntary Contraction (MVC). In addition, the timing of each muscle activiation during gait cycle will be extracted to compared before and after training. This includes identifying the onset (activation start) and offset (activation end) of each muscle relative to specific phases of the gait cycle, such as the stance and swing phases.
Fugl-Meyer assessment (FMA-LE) | At baseline and 6 weeks post-intervention
  The lower extremity motor subscale of the Fugl-Meyer assessment (FMA-LE) was used to measure the level of lower extremity motor recovery after stroke. Quality of reflexes, coordination and voluntary movements of the paretic leg was assessed using a 0-to-34-point scale. Higher FMA-LE score indicated a better level of motor recovery.
Berg Balance Scale (BBS) | At baseline and 6 weeks post-intervention
  Berg Balance Scale (BBS) was adopted to measure functional balance performance. The scale consists of 14 items, each rating a participant's ability to maintain stability in a specified functional task on a 5 point (0-4) scale. The maximal score of BBS is 56 and minimum is 0, with a higher score indicating better balance performance.
Subjective Index of physical and Social Outcome (SIPSO) | At baseline and 6 weeks post-intervention
  The Chinese version of the subjective Index of physical and Social Outcome (SIPSO) questionnaire assesses the extent to which individuals with disabilities are able to function physically and socially to their own satisfaction. It is a 5 point (0-4) scale, the maximal score of SIPSO is 40 and minimum score is 0, with a higher score indicating better physical and social integration.
Short Physical Performance Battery (SPPB) | At baseline and 6 weeks post-intervention
  The Short Physical Performance Battery (SPPB) is a tool used to assess lower extremity function and physical performance in older adults. It includes three components:
  Balance Tests: Measures ability to maintain balance in different stances. Gait Speed: Assesses walking speed over a short distance. Chair Stand Test: Evaluates leg strength by timing how quickly one can stand from a seated position multiple times.
  The maximum score is 12 and the minimum score is 0, a higher score indicates better physical performance and functional ability.
Trunk Impairment Scale (TIS) | At baseline and 6 weeks post-intervention
  The Trunk Impairment Scale (TIS) is an assessment tool used to evaluate trunk control and stability. It is primarily used for individuals with neurological conditions, such as stroke. The scale measures:
  Static Sitting Balance: Ability to maintain a stable sitting position. Dynamic Sitting Balance: Ability to maintain balance while moving. Coordination: Assesses coordinated trunk movements. It has a maximum score of 23 and minimum score of 0. The higher the score, the better the trunk control, stability, and coordination.
Ability to Perform Locomotion Activities (ABILOCO) | At baseline and 6 weeks post-intervention
  ABILOCO is a questionnaire designed to assess locomotion and daily-life ability in individuals. It evaluates a person's capacity to perform various mobility tasks, ranging from simple to complex. The ABILOCO scale typically ranges from a minimum score of 0 to a maximum score of 59, where higher scores indicate better locomotion ability and greater independence in performing mobility tasks.
Timed Up and Go (TUG) test | At baseline and 6 weeks post-intervention
  The Timed Up and Go (TUG) test was used to assess functional mobility, balance, and fall risk. Participants were instructed to stand up from a standard chair (45cm-height), walk a distance of 3 meters, turn around, walk back to the chair, and sit down. The total time taken to complete the task was recorded in seconds using a stopwatch. A shorter completion time indicates better functional mobility, while longer times may reflect impaired mobility or increased fall risk.

CONTACTS AND LOCATIONS:
Locations (1):
- the Hong Kong Polytechnic University, Hksar, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to other researchers